CLINICAL TRIAL: NCT05523063
Title: Effects on Quality of Life of Adapted Physical Activity Supervised by CAMI for Breast Cancer Patients.
Brief Title: Effect of Physical Activity in Patients With Breast Cancer.
Acronym: APACAM
Status: Withdrawn | Type: Observational
Why Stopped: Study classified as out of scope by the Ethics Committee (not a project involving human person).
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL22_0613
Record Dates: First submitted 2022-08-29; First posted 2022-08-31 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Breast Cancer
Keywords: Adapted physical activity; Quality of life; Breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Breast cancer patients followed at CAMI: The trial population concerns all adult patients with breast cancer followed at the Croix-Rousse hospital, who have been under care for less than 3 months or who are going to be treated at the CAMI.
  Interventions: Other: Quality of life questionnaire

INTERVENTIONS:
Other: Quality of life questionnaire — The quality of life questionnaire will be performed in routine practice by the CAMI during the initial assessment.
  The 3-month visit is part of the routine patient visit to CAMI. During this visit, the quality of life questionnaire will be completed a second time by the patients, through a phone call given by the investigator.

SUMMARY:
Every year in France, there are approximately 58,000 new cases of breast cancer, which is the leading cancer in women according to the National Cancer Institute.

Among the various tools in the fight against cancer, it is now proven that physical activity improves the prognosis of cancers, particularly breast cancer.

Indeed, APA (Adapted Physical Activity) reduces morbidity and mortality, the risk of recurrence and improves quality of life. It is one of the tools of the Ten-Year Cancer Control Strategy 2021-2030 of the anti-cancer plan.

However, it seems to be insufficiently proposed and prescribed in France at present.

CAMI (Cancer Arts Martiaux et Information) is a non-profit association comprising health professionals specifically trained to support cancer patients through APA. It works in collaboration with the Hospices Civils de Lyon and in particular the Gynecology Department of the CHU (University Hospital Center) of Croix Rousse.

According to the World Health Organization (WHO), quality of life is "an individual's perception of his or her place in life, in the context of the culture and value system in which he or she lives, in relation to his or her goals, expectations, norms and concerns. It is a very broad concept influenced in a complex way by the subject's physical health, psychological state, level of independence, social relationships as well as their relationship to the essential elements of their environment."

Quality of life is thus synonymous with well-being, perceived health and life satisfaction. The quality of a person's life is based both on the objective elements of his or her life (physical health, living environment and material and/or contextual conditions) and on his or her experience, which can be defined as the subjective quality of life.

Thus, quality of life is considered to be a multidimensional concept that is structured around four dimensions, the first of which encompasses the physical state (autonomy, physical abilities), the second the somatic sensations that often translate into the expression of pain, the consequences of trauma related to the disease or treatment.

With the increase in the incidence of breast cancer and the improvement in its prognosis, the number of breast cancer survivors has increased significantly. Quality of life has become an important outcome measure in clinical breast cancer surveys and survival studies, in addition to survival.

The investigators' main objective is to study the effects of APA managed by CAMI in routine practice, on the quality of life of breast cancer patients.

They also want to analyze how, by whom, and which patients are referred to CAMI to improve their care and describe the program offered by CAMI.

The aim of this research is therefore to establish an axis of work and improvement for the Gynecology Department of the Croix Rousse Hospital in order to better identify the patients for whom APA would be most beneficial, to better refer them to CAMI and to study in real practice the effects of APA on these patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years or older at inclusion,
* With breast cancer (diagnosis of breast cancer proven by anatomopathological evidence; all stages of the disease accepted), including recurrences,
* Followed at the Croix-Rousse Hospital and managed by the CAMI for less than 3 months,
* Provision of an informed information and collection of non-opposition.

Exclusion Criteria:

* Patients who do not speak French,
* Persons of legal age who are the subject of a legal protection measure,
* Persons deprived of liberty by a judicial or administrative decision, persons under psychiatric care,
* Pregnant or parturient women.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The trial population concerns all adult patients with breast cancer followed at the Croix-Rousse hospital, who have been under care for less than 3 months at CAMI or who are going to be treated at CAMI.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Change in Quality of life questionnaire score | Change from Baseline Score of the Quality of life at 3 months
  Difference between the quality of life questionnaire score calculated at baseline (first visit at CAMI) and after 3 months of follow-up by CAMI. The minimum and maximum values of the Quality of life questionnaire are respectively 0 (bad quality of life) and 100 (good quality of life).

CONTACTS AND LOCATIONS:
Overall Officials: Marion CORTET, MD, Principal Investigator — Service de Gynécologie-Obstétrique, Hôpital de la Croix-Rousse, Hospices Civils de Lyon
Locations (1):
- Service de Gynécologie-Obstétrique, Hôpital de la Croix-Rousse, Hospices Civils de Lyon, Lyon, France